CLINICAL TRIAL: NCT06900920
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQB3473 Tablets Compared to Placebo in the Treatment of Adult Primary Immune Thrombocytopenia (ITP)
Brief Title: A Study of TQB3473 Tablets Compared to Placebo in the Treatment of Adult Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB3473-III-01
Record Dates: First submitted 2025-03-24; First posted 2025-03-28 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-11

CONDITIONS: Primary Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQB3473 Tablets (Active Comparator): TQB3473 Tablets 600 mg orally once daily for 24 consecutive weeks.
  Interventions: Drug: TQB3473 Tablets
- TQB3473 Placebo (Placebo Comparator): Placebo, orally once daily for 24 consecutive weeks.
  Interventions: Drug: TQB3473 Placebo

INTERVENTIONS:
Drug: TQB3473 Tablets — TQB3473 tablet is a selective Spleen tyrosine kinase (Syk) inhibitor.
  Arms: TQB3473 Tablets
Drug: TQB3473 Placebo — Placebo contains no active substance.
  Arms: TQB3473 Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled Phase III clinical study designed to demonstrate that TQB3473 tablets significantly improve the sustained response rate compared to placebo in adult patients with chronic ITP who have previously received standard corticosteroid therapy and have failed or relapsed after at least one standard ITP treatment.

The study consists of a treatment period and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily join this study, sign the informed consent form (ICF), and demonstrate good compliance;
* Male or female subjects aged 18 to 75 years (calculated based on the date of signing the informed consent form);
* Eastern Cooperative Oncology Group (ECOG) score of 0-1;
* Diagnosis of primary ITP prior to randomization, with a duration of ≥12 months;
* An average of at least three independent platelet counts (spaced more than 3 days apart) within the 3 months prior to randomization <30×10^9/L, with no count >35×10^9/L; and no severe bleeding within 4 weeks prior to screening;
* Previous treatment with glucocorticoids and at least one standard ITP therapy that was ineffective or resulted in relapse.
* Female subjects of childbearing potential must agree to use effective contraception during the study and for 6 months after the end of study treatment, with a negative serum or urine pregnancy test within 7 days prior to study enrollment; male subjects must agree to use effective contraception during the study and for 6 months after the end of study treatment, as detailed in Section 5.5.

Exclusion Criteria:

* Evidence of secondary causes of ITP (e.g., untreated Helicobacter pylori infection, leukemia, lymphoma, history of autoimmune diseases such as systemic lupus erythematosus, Hashimoto's thyroiditis, etc.) or drug-induced causes (e.g., anticonvulsants, antibiotics, heparin, etc.), or immune-mediated cytopenia involving two or more cell lines such as Evans syndrome or immune-related cytopenia;
* Subjects with a history or current diagnosis of myelofibrosis, myelodysplastic syndrome, aplastic anemia, lymphoproliferative disorders, or other malignant hematologic diseases;
* History of or concurrent other malignancies within the past 3 years. Exceptions include: other malignancies treated with a single surgical procedure and achieving continuous 5-year disease-free survival (DFS); cured cervical carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor invading the basement membrane)];
* Conditions affecting venous blood sampling or multiple factors affecting oral medication (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.);
* Adverse reactions from previous treatments have not resolved to ≤CTCAE grade 1, except for non-clinically significant and asymptomatic laboratory abnormalities judged by the investigator to pose no safety risks;
* Previous bone marrow/hematopoietic stem cell transplantation or major solid organ transplantation;
* Vaccination within 8 weeks prior to randomization or planned vaccination during the study period;
* Major surgical treatment or significant traumatic injury within 4 weeks prior to randomization, or anticipated need for major elective surgery during the study treatment period (major surgery is defined as level 3 or higher according to the National Surgical Classification Catalog 2022);
* History of intracranial hemorrhage or other severe bleeding in vital organs (≥CTCAE grade 3), or symptomatic gastrointestinal bleeding (e.g., hematemesis, melena, etc., excluding asymptomatic "occult blood test positive" and hemorrhoids) within 6 months prior to screening;
* Arterial/venous thrombotic events within 12 months prior to randomization, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism;
* ITP-related symptoms and treatments:

  1. Receipt of immunoglobulins or platelet transfusions within 2 weeks prior to randomization;
  2. Receipt of treatments aimed at increasing platelet counts (including but not limited to glucocorticoids, Thyroid peroxidase (TPO), Thrombopoietin receptor agonists (TPO-RAs), cyclosporine, herbal medicines, etc.) within 4 weeks prior to randomization, except for those meeting inclusion criterion (8);
  3. Use of rituximab or other anti-cluster of differentiation 20 (CD20) drugs within 14 weeks prior to randomization;
  4. Splenectomy within 12 weeks prior to randomization.
* Need for long-term/continuous use of medications affecting platelet function [including but not limited to aspirin, clopidogrel, ticagrelor, non-steroidal anti-inflammatory drugs (NSAIDs), etc.] or anticoagulant therapy;
* Known allergy to the active ingredient or excipients of the investigational drug;
* Previous treatment with Syk inhibitors;
* Participation in another clinical trial and use of investigational drugs within 4 weeks prior to randomization;
* Any condition judged by the investigator to pose a significant risk to the subject's safety or to affect the subject's ability to complete the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Durable response rate: platelet counts ≥50×10^9/L | During the 24-week randomized double-blind treatment period (Weeks 14-24)
  During the 24-week randomized double-blind treatment period (Weeks 14-24), platelet counts ≥50×10^9/L in at least 4 out of the 6 protocol-specified visits (excluding rescue treatment).

SECONDARY OUTCOMES:
The effectiveness rate within the first 12 weeks of treatment | Baseline to 12 weeks
  ①The proportion of subjects with at least one platelet count ≥50×10^9/L during weeks 1-12 (excluding emergency treatment).②Among subjects with a baseline platelet count <15×10^9/L, the proportion of subjects with at least one platelet count ≥30×10^9/L and an increase of ≥20×10^9/L from baseline during weeks 1-12 (excluding rescue treatment).
The response rate within 24 weeks of treatment | 24 weeks
  ① The proportion of subjects with at least one platelet count ≥50×10^9/L during weeks 1-24 (excluding rescue treatment).
  ② Among subjects with a baseline platelet count <15×10^9/L, the proportion of subjects with at least one platelet count ≥30×10^9/L and an increase of ≥20×10^9/L from baseline during weeks 1-24 (excluding rescue treatment).
  ③ The proportion of subjects with platelet counts at least twice the baseline level and ≥30×10^9/L for at least two consecutive measurements during weeks 1-24 (excluding rescue treatment).
Time to response: The time from the initiation of treatment to the first platelet count ≥50×10^9/L | The time from the initiation of treatment to the first platelet count ≥50×10^9/L (excluding rescue treatment)
  The time from the initiation of treatment to the first platelet count ≥50×10^9/L
The incidence and severity of bleeding events (Weeks 1-12) | During Weeks 1-12 of the double-blind treatment period
  During Weeks 1-12 of the double-blind treatment period, the incidence and severity of bleeding events as assessed by the World Health Organization (WHO) bleeding score.
The incidence and severity of bleeding events (Weeks 1-24) | During Weeks 1-24 of the double-blind treatment period
  During Weeks 1-24 of the double-blind treatment period, the incidence and severity of bleeding events as assessed by the World Health Organization (WHO) bleeding score.
The proportion of subjects who receive rescue treatment | During the 24-week double-blind treatment period
  The proportion of subjects who receive rescue treatment aimed to increase platelet counts during the 24-week double-blind treatment period.
The change of concomitant therapy | During the 24-week double-blind treatment period
  The proportion of subjects who reduce or discontinue concomitant ITP treatments during the 24-week double-blind treatment period.
The incidence and severity of adverse events | From the signing of the informed consent until 28 days after the last dose of study drug or the initiation of new ITP treatment, whichever occurs first
  The proportion of subjects experiencing adverse events and the severity of these events, with adverse events assessed using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Locations (53):
- China (53):
  - The first affiliated hospital of ustc anhui provincial hospital, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Nanshan People's Hospital, Shenzhen, Guangdong
  - Central People's Hospital of Zhanjiang, Zhanjiang, Guangdong
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The First Affiliated Hospital of Hainan Medical University, Haikou, Hainan
  - Affiliated Hospital of Hebei University / School of Clinical Medicine, Baoding, Hebei
  - Affiliated Hospital of ChengDe Medical University, Chengde, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - North China University of science and technology, Tangshan, Hebei
  - The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Anyang People's Hospital, Anyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Xuchang Central Hospital, Xuchang, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First People's Hospital of Ping Ding Shan, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The Third Hospital of Changsha, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Northern Jiangsu People's Hospital Affiliated to Yangzhou University, Yangzhou, Jiangsu
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - Shenjing Hospital Of China Medical University, Shenyang, Liaoning
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Xijing Hospital, Xi'an, Shaanxi
  - Xi'an No.3 Hospital, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong First Medical University Affiliated Central Hospital, Jinan, Shandong
  - Linyi Central Hospital, Linyi, Shandong
  - Yantai Yuhuangding Hospital (Affiliated Yantai Yuhuangding Hospital of Qingdao University), Yantai, Shandong
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University，Qingpu Branch, Shanghai, Shanghai Municipality
  - Heping Hospital affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Kunming Medical University Second Affiliated Hospital, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang